CLINICAL TRIAL: NCT00956631
Title: MiDAS I (Mild® Decompression Alternative to Open Surgery): Vertos Mild Patient Evaluation Study
Acronym: MiDAS I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vertos Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MiDAS I
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-02

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Spinal Stenosis; Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- interlaminar decompression (Other): Commercially available product (mild® Device Kit) used to perform interlaminar decompression
  Interventions: Procedure: Interlaminar Decompression

INTERVENTIONS:
Procedure: Interlaminar Decompression — The MILD® devices used in this study are specialized surgical instruments intended to be used to perform percutaneous lumbar decompression.
  Other Names: mild® Device Kit; percutaneous decompression

SUMMARY:
This is a multi-center, prospective, clinical study to assess the clinical application and outcomes of MILD® Interlaminar Decompression in patients with symptomatic lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Lumbar Spinal Stenosis (LSS) primarily caused by dorsal element hypertrophy.
* Prior failure of conservative therapy.
* Radiologic evidence of LSS (L3-L5), Ligamentum flavum > 2.5mm, confirmed by pre-op MRI and/or CT.
* Central canal cross sectional area ≤ 100 square mm.
* Anterior listhesis ≤ 5.0mm.
* Able to walk at least 10 feet unaided before being limited by pain.
* Available to complete 12 weeks of follow-up.
* Consistent with the intended labeling statement for use.
* Able to use all package components to perform the procedure.
* A signed Informed Consent Form is obtained from the patient.

Exclusion Criteria:

* Prior surgery at intended treatment level.
* History of recent spinal fractures with concurrent pain symptoms.
* Disabling back or leg pain from causes other than LSS (e.g. acute compression fracture, metabolic neuropathy, or vascular claudication symptoms, etc.).
* Significant / symptomatic disk protrusion or osteophyte formation.
* Excessive / symptomatic facet hypertrophy.
* Bleeding disorders and/or current use of anti-coagulants.
* Use of acetylsalicylic acid (ASA) and/or non-steroidal anti-inflammatory drug (NSAID) within 5 days of treatment.
* Epidural steroids within prior three weeks.
* Inability of the patient to lie prone for any reason with anesthesia support (e.g. chronic obstructive pulmonary disease (COPD), obesity, etc.).
* Any potential wound healing pathologies that may compromise outcomes, including diabetes, excessive smoking history, cancer, connective tissue diseases, recent spine radiation and severe COPD.
* Dementia and/or inability to give informed consent.
* Pregnancy.
* Intended treatment that is defined by the product labeling contraindications.
* On Workman's Compensation or considering litigation associated with back pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Caraway, MD, Principal Investigator — The Center for Pain Relief Tri-State, PLLC; Bohdan W Chopko, MD, Principal Investigator — MedCentral Health System
Locations (13):
- United States (13):
  - NEA Clinic, Jonesboro, Arkansas
  - UCLA, Los Angeles, California
  - Napa Pain Institute, Napa, California
  - Scripps, Division of Orthopedic Surgery, San Diego, California
  - UCSD, San Diego, California
  - Your Pain Care, Temecula, California
  - Coastal Orthopedics & Sports Medicine, Bradenton, Florida
  - South Florida Spine Institute, Miami Beach, Florida
  - The Spine Center, Baltimore, Maryland
  - Rainer Vogel, MD LTD, Henderson, Nevada
  - Lab2Marche, LLC, Las Vegas, Nevada
  - MedCentral Health System, Mansfield, Ohio
  - Orthopedic Associates of the Greater Lehigh Valley, Easton, Pennsylvania

REFERENCES:
- [Derived] Chopko B, Caraway DL. MiDAS I (mild Decompression Alternative to Open Surgery): a preliminary report of a prospective, multi-center clinical study. Pain Physician. 2010 Jul-Aug;13(4):369-78. PMID 20648206

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient enrollment July 2008 to January 2010 at fourteen study sites. Treatments were performed in an outpatient setting at an hospital outpatient or ambulatory surgery center.
Pre-assignment Details: After enrollment and prior to surgery patient was excluded if patient had procedure or trauma at study treatment level, used acetylsalicylic acid (ASA) or non-steroidal anti-inflammatory drug (NSAID) within five days of treatment, epidural steroid injection (ESI) within 3 weeks of treatment.
Groups:
- Mild Procedure: Symptomatic lumbar spinal stenosis (LSS) patients having neurogenic claudication complaints and predominant causal factor of hypertrophic ligamentum flavum were treated with the mild® device kit in a percutaneous decompression procedure.
Period: Overall Study
Arm/Group | Mild Procedure
Started | 78
Completed | 62
Not Completed | 16

BASELINE CHARACTERISTICS:
Groups:
- Mild Procedure: Symptomatic LSS patients having neurogenic claudication complaints and predominant causal factor of hypertrophic ligamentum flavum were treated with the mild® device kit in a percutaneous decompression procedure.
Arm/Group | Mild Procedure
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 70 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Back Pain as Measured by a 10-point Visual Analog Scale (VAS).
Description: The 10-point Visual Analog Scale rates 'no pain' as zero and 'worst pain imaginable' as ten. Visual analog scores of mean improvement greater than or equal to 2.0 are clinically relevant. The change from baseline to six months is reported below, where a positive value represents the baseline value minus the 6 month value.
Time Frame: Baseline and Six Months
Population: All available treated patients at Month 6.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mild Procedure: Percutaneous decompression with the mild device kit.
Arm/Group | Mild Procedure
Number analyzed (Participants) | 62
units on a scale | 3.21 (p<0.0001) [2.29 to 4.13]
Statistical Analysis 1: Comparison: Mild Procedure; The mean change from baseline was assessed for VAS using a paired t-test. The resulting p-values are to be considered as descriptive statistics. Two-sided test with 5% Type I error was used throughout. A hypothetical average improvement of zero was used; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [2.29 to 4.13]

2. Other Pre Specified Outcome: Function Measure Oswestry Disability Index (ODI). Measures Permanent Functional Disability Through Questions Which Characterize Disturbance of Activities of Daily Living (ADL) Resulting From Chronic Back Pain. Higher Scores Indicate Greater Disability.
Description: Change from baseline to month six is reported below, where a positive value represents baseline value minus 6 month value. The questionnaire is divided into 10 topics including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling and employment/homemaking. Each topic is rated 0 (no pain or no limitation)to 5 (high pain or very limited physically) based on typical pain and/or physical limitations. The worst possible score is 50 (100 % disability) and best would be zero (0% disability).
Time Frame: Baseline and Six months
Population: All available participants at Month 6.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mild Procedure: Percutaneous lumbar decompression with the mild device kit.
Arm/Group | Mild Procedure
Number analyzed (Participants) | 62
units on a scale | 17.58 [12.33 to 22.83]
Statistical Analysis 1: Comparison: Mild Procedure; The mean change from baseline was assessed for ODI using a paired t-test. The resulting p-values are to be considered as descriptive statistics. Two-sided test with 5% Type I error was used. A hypothetical average improvement of zero was used; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 17.58, 95% CI 2-sided [12.33 to 22.83]

3. Other Pre Specified Outcome: Quality of Life Physical Component Score (PCS) as Measured by the 12-question Short Form Survey Version 2 (SF-12v2). Change From Baseline Mean to Six Month Mean is Reported Below. A Positive Value Represents the 6 Month Value Minus the Baseline Value.
Description: Minimally Important Difference (MID) is a measure of true clinical relevance of a difference. The MID for mean Physical Component Score (PCS) improvement is 2 to 3 points. SF-12v2 is a validated tool that uses norm-based scoring to determine treatment outcomes & is a generic measure, as opposed to one that targets a specific age, disease, or treatment group. The SF-12v2 asks for patient views about their health to determine how they feel & how well they are able to conduct their usual activities. The data for the 2 summary scales and 8 survey scales are normalized so each scale has the same mean (50 points) & the same standard deviation (10 points) in the general 1998 U.S. population. By using this method, anytime a scale is below 50, health status is below average, & each point is one-tenth of a standard deviation. The PCS summary measure takes into account the correlations among the Health Survey scales, & shows the broad impact which was of interest in this study.
Time Frame: Baseline and Six Months
Population: All available participants were analyzed at six months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mild Procedure: Symptomatic lumbar spinal stenosis (LSS) patients having neurogenic claudication complaints and predominant causal factor of hypertrophic ligamentum flavum were treated using the mild® device kit in a percutaneous lumbar decompression procedure.
Arm/Group | Mild Procedure
Number analyzed (Participants) | 62
units on a scale | 7.11 (11.32) [3.62 to 10.60]

ADVERSE EVENTS:
Arm/Group | Mild Procedure
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less